CLINICAL TRIAL: NCT03825133
Title: The Comparison of Knee Osteoarthritis Treatment With Single-dose of Bone Marrow Aspirate Concentrate, Single-dose of Leukocyte Rich Platelet Rich Plasma and 3 Injection of High Molecular Weight Hyaluronic Acid-A Randomized Clinical Trial
Brief Title: The Comparison of Knee Osteoarthritis Treatment With Bone Marrow Aspirate Concentrate , Leukocyte Rich Platelet Rich Plasma and Hyaluronic Acid
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Clinical Center of Vojvodina (Other)
Responsible Party: Principal Investigator, dr Oliver Dulic, Oliver Dulic MD, M.sci . Orthopaedic Surgeon, Principal Investigator, Clinical Center of Vojvodina
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CCVBMACKnee
Record Dates: First submitted 2019-01-23; First posted 2019-01-31 (Actual); Last update posted 2019-02-07 (Actual); Status verified 2019-02

CONDITIONS: Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Hyaluronic Acid

STUDY DESIGN:
Intervention Model Description: Patients will be randomly assigned to 3 groups: LR-PRP group, the BMAC group or HA group. Functional scores and outcomes will be compared to determine clinical efficacy of all groups and which treatment is more effective in treating knee OA
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Bone Marrow Aspirate Concentrate (Experimental): Patients treated with single injection of BMAC in the knee
  Interventions: Procedure: Bone Marrow Aspirate Concentrate
- Leukocyte Rich Platelet Rich Plasma (Experimental): Patients treated with single injection of LR-PRP in the knee
  Interventions: Procedure: Leukocyte Rich Platelet Rich Plasma
- Hyaluronic Acid (Experimental): Patients treated with 3 single injection of high molecular HA in the knee ( one injection weekly)
  Interventions: Drug: Hyaluronic Acid

INTERVENTIONS:
Procedure: Bone Marrow Aspirate Concentrate — Bone marrow ( 100 ml) is aspirated from proximal tibia, concentrated in Arthrex Angel Centrifuge, and after concentration 6 ml of BMAC is injected in the knee
  Other Names: BMAC
  Arms: Bone Marrow Aspirate Concentrate
Procedure: Leukocyte Rich Platelet Rich Plasma — Blood sample is taken ( 100 ml), centrifuged in Arthrex Angel Centrifuge and after double spinning process about 6 ml of PRP is injected in the knee
  Other Names: LR-PRP
  Arms: Leukocyte Rich Platelet Rich Plasma
Drug: Hyaluronic Acid — Three injections of Cartinorm (1% Sodium Hyaluronat (20mg/2 ml) by Goodwill Pharma) is injected in the knee weekly
  Other Names: HA
  Arms: Hyaluronic Acid

SUMMARY:
The aim of this study is to compare therapeutic and clinical effects of intra-articular injection of Bone Marrow Aspirate Concentrate (BMAC), inta-articular injection of Leukocyte Rich Platelet Rich plasma (LR-PRP) and 3 weekly doses of high molecular weight of Hyaluronic acid for the treatment of osteoarthritis (OA) of the knee ( KL scale II-IV).

DETAILED DESCRIPTION:
Osteoarthritis (OA) is the most common joint disease worldwide, affecting an estimated 10% of men and 18% of women over 60 years of age with the knee and hip joints predominantly involved. The pain and loss of function can be debilitating; in developed countries the resultant socioeconomic burden is large costing between 1, 0% and 2, 5% of gross domestic product. Several therapeutic options for the treatment of OA are widely used, consists of pain management, physical therapy with life-modifying recommendations, joint injections with joint replacement for end-stage disease. Intra-articular drug delivery has several advantages over systemic delivery, including increased local bioavailability, reduced systemic exposure, fewer adverse events and reduced cost. Three injectable materials have been widely used for intra-articular treatment of the knee OA: corticosteroids (with or without local anesthetics), hyaluronic acid based preparations and in the last decade biologic preparations, such as human serum albumin, TNF and Il-1 inhibitors, platelet-rich plasma (PRP) injections, bone marrow-derived stem cells (BMSCs), adipose-derived stem cells (ADSCs) and amnion-derived mesenchymal stem cells (AMSCs) etc PRP is promising therapeutic option for the OA treatment, there are still many concerns with PRP's efficiency. Among all questions, ( Number of platelets, percentage in accordance with baseline, frequency of doses etc.) presence or absence of different cells in PRP formulations ( as leukocytes), could significantly change an overall clinical result. In general, PRP could be Leukocyte-rich (LR- with increase number of Leukocytes in comparison with baseline number) and Leukocyte-poor.

Another option that has become more popular for physicians treating this debilitation condition is BMAC, which use undifferentiated cells found in the bone marrow to promote healing and tissue regeneration. These cells have the ability to replicate into a multiple different tissue types. With BMAC, the marrow is concentrated provide better healing of the damaged tissue and aid in growth and repair. The full benefits of BMAC are still unknown, but studies have shown the treatment can reduce swelling, relieve pain, and improve healing in articular cartilage and bone grafts.

Autologous BMAC has shown promising clinical potential as a therapeutic agent in regenerative medicine, including the treatment of osteoarthritis and cartilage defects, and the clinical efficacy platelet rich plasma has been documented to alleviate symptoms related to knee osteoarthritis. However, randomized, prospective comparison of the two techniques has not been reported in the literature and long term follow-up for both treatments is limited, and especially limited in the use of BMAC for the knee OA treatment.

From the other hand, HA preparations are widely used in everyday practice for almost 30 years with variable results. No one of these therapeutic options are not yet recommended by supreme professional organizations ( e.g.AAOS) because of paulacity of scientific data and unbiased confirmation of their clinical efficiency with a broad advice for necessity of more rigorous clinical trials.

ELIGIBILITY:
Inclusion Criteria:

* history of complaints of knee pain because of the Knee Osteoarthritis with no relief using anti-inflammatory agents even after 3 months,
* Kellgren-Lawrence (KL) grade 2-4
* normal blood results and coagulation profile (platelets 150,000-450,000/l),
* patients who had not undergone any surgery on the affected knee within 2 years prior to the first injection and
* Mentally fit for clinical study

Exclusion Criteria:

* severe knee instability,
* severe misalignment,
* unicompartmental OA
* BMI more than 35
* inflammatory arthritis such as rheumatoid arthritis and ankylosing spondylitis
* presenting muscle pain underlying diseases such as hematologic disorders, septicemia, coagulopathy, neoplasm, active infection, and immune deficiency

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2016-04-01 (Actual); Primary Completion 2017-11-30 (Actual); Study Completion 2017-11-30 (Actual)

PRIMARY OUTCOMES:
change of WOMAC | after 1, 3, 6, 9 and 12 months
  Purpose of WOMAC scale is to assess the course of disease or response to treatment in patients with knee or hip osteoarthritis (OA).Content: Three subscales, 24 items.: 1) pain severity during various positions or movements, 2) severity of joint stiffness, and 3) difficulty performing daily functional activities.Response options/scale: In the Likert version, each item offers 5 responses: "none" scored as 0, "mild" as 1,"moderate" as 2, "severe" as 3, and "extreme" as 4. Alternatively, the VAS and numerical rating scale versions permit responses to be selected on a 100-mm or 11-box horizontal scale, respectively, with the left end marked as "none" and the right end marked as "extreme". The range for possible subscale scores in the Likert format are: pain (0-20; 5 items each scored 0-4), stiffness (2 items, 0-8), and physical function (17 items, 0-68). Score interpretation: Higher scores indicate worse pain, stiffness, or physical function.
Change of KOOS | after 1, 3, 6, 9 and 12 months
  Purpose of KOOS is To measure patients' opinions about their knee and associated problems over short- and long-term follow- up Intended populations/conditions: young and middle-aged people with posttraumatic osteoarthritis (OA), as well as those with injuries that may lead to post traumatic OA (e.g., ACL, meniscal, osteochondral injury) Content. Five domains: 1) pain frequency and severity during functional activities; 2) symptoms such as the severity of knee stiffness and the presence of swelling, grinding or clicking, catching, and range of motion restriction; 3) difficulty experienced during activities of daily living; 4) difficulty experienced with sport and recreational activities; and 5) knee-related quality of life.Number of items: 42 items across 5 subscales.
  Score interpretation: 0- extreme problems and 100- no problems.

SECONDARY OUTCOMES:
change of SF-36 | after 1, 3, 6, 9 and 12 months
  The SF-36 is multi-item generic health surveys intended to measure "general health concepts not specific to any age, disease, or treatment group" . The original objective was to develop a short, generic health-status measure that reproduces the 2 summary scores of the SF-36, i.e., the physical component summary (PCS) score and the mental component summary (MCS) score (2).
  The SF-36 consists of 36 items, 35 of which are used in the calculation of 8 separate scale scores. The physical functioning scale (10 items) is the longest scale.
  Scores on the SF-36 and SF-12 scales range from 0-100, with higher scores indicating better health. On the physical functioning scale, low scores are typical of someone who experiences many limitations in physical activities, including bathing or dressing, while high scores represent someone who is able to perform these types of activities without limitations
Change of IKDC | after 1, 3, 6, 9 and 12 months
  Purpose of IKDC is to detect improvement or deterioration in symptoms, function, and sports activities due to knee impairment Intended populations/conditions: Patients with a variety of knee conditions, including ligament injuries, meniscal injuries, articular cartilage lesions, and patellofemoral pain.
  Content: Three domains: 1) symptoms, including pain, stiffness, swelling, locking/catching, and giving way; 2) sports and daily activities; and 3) current knee function and knee function prior to knee injury (not included in the total score).
  Number of items.18 (7 items for symptoms, 1 item for sport participation, 9 items for daily activities, and 1 item for current knee function).
  Possible score range 0-100, where 100 means no limitation with daily or sporting activities and the absence of symptoms.
change of VAS pain | after 3, 7 14 and 21 days
  The pain VAS is a unidimensional measure of pain intensity, which has been widely used in diverse adult populations, including those with rheumatic diseases .The pain VAS is a continuous scale comprised of a horizontal (HVAS) or vertical (VVAS) line, usually 10 centimeters (100 mm) in length, anchored by 2 verbal descriptors, one for each symptom extreme. Instructions, time period for reporting, and verbal descriptor anchors have varied widely in the literature depending on intended use of the scale.The pain VAS is a single-item scale. For pain intensity, the scale is most commonly anchored by "no pain" (score of 0) and "pain as bad as it could be" or "worst imaginable pain" (score of 100 [100-mm scale]) (6-8). To avoid clustering of scores around a preferred numeric value, numbers or verbal descriptors at intermediate points are not recommended .A higher score indicates greater pain intensity.
VAS pain injection | up to 10 minutes after after intervention
  The pain VAS is a unidimensional measure of pain intensity, which has been widely used in diverse adult populations, including those with rheumatic diseases .The pain VAS is a continuous scale comprised of a horizontal (HVAS) or vertical (VVAS) line, usually 10 centimeters (100 mm) in length, anchored by 2 verbal descriptors, one for each symptom extreme. Instructions, time period for reporting, and verbal descriptor anchors have varied widely in the literature depending on intended use of the scale.The pain VAS is a single-item scale. For pain intensity, the scale is most commonly anchored by "no pain" (score of 0) and "pain as bad as it could be" or "worst imaginable pain" (score of 100 [100-mm scale]) (6-8). To avoid clustering of scores around a preferred numeric value, numbers or verbal descriptors at intermediate points are not recommended .A higher score indicates greater pain intensity.
VAS score after injection of fluid | up to 10 minutes after after intervention
  The pain VAS is a unidimensional measure of pain intensity, which has been widely used in diverse adult populations, including those with rheumatic diseases .The pain VAS is a continuous scale comprised of a horizontal (HVAS) or vertical (VVAS) line, usually 10 centimeters (100 mm) in length, anchored by 2 verbal descriptors, one for each symptom extreme. Instructions, time period for reporting, and verbal descriptor anchors have varied widely in the literature depending on intended use of the scale.The pain VAS is a single-item scale. For pain intensity, the scale is most commonly anchored by "no pain" (score of 0) and "pain as bad as it could be" or "worst imaginable pain" (score of 100 [100-mm scale]) (6-8). To avoid clustering of scores around a preferred numeric value, numbers or verbal descriptors at intermediate points are not recommended .A higher score indicates greater pain intensity.

OTHER OUTCOMES:
Knee injection portals influence on final clinical results. | after one year
  We used three most widely used portals: (1) The anterolateral portal (AL) where patient is supine, with a knee in full extension where a needle is placed 1 cm above the joint line and just next to the patellar tendon in a palpable soft spot with the knee passively fully flexed to a tolerable degree for the patient ranging from 100 to 130, with a foot internally rotated. (2) The anteromedial portal (AM) is placed 1 cm above the joint line and 1 cm medial to the patellar tendon, also in a palpable soft and (3) Superolateral portal ( SL) involved insertion of a needle 1 cm above and 1 cm lateral to the superior lateral aspect to the patella at a 45 degrees angle. Then, patients were asked to describe pain during injection procedure alone using Visual Analog Scale After 12 months, we calculate, are there any statistical differences in previous scales ( WOMAC, KOOS, IKDC, SF-26) in accordance with a portal placement.

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Center of Vojvodina, Novi Sad, Vojvodina, Serbia

IPD SHARING:
Plan to Share IPD: Yes
de-identified individual participant data for all primary and secondary outcome measures will be made available.
Supporting Information: SAP, ICF, CSR
Time Frame: after data analyze

REFERENCES:
- [Background] Chahla J, Alland JA, Verma NN. Bone Marrow Aspirate Concentrate for Orthopaedic Use. Orthop Nurs. 2018 Nov/Dec;37(6):379-381. doi: 10.1097/NOR.0000000000000502. PMID 30451775
- [Background] Chahla J, Mandelbaum BR. Biological Treatment for Osteoarthritis of the Knee: Moving from Bench to Bedside-Current Practical Concepts. Arthroscopy. 2018 May;34(5):1719-1729. doi: 10.1016/j.arthro.2018.01.048. Epub 2018 Apr 5. PMID 29628381
- [Background] Jones IA, Togashi R, Wilson ML, Heckmann N, Vangsness CT Jr. Intra-articular treatment options for knee osteoarthritis. Nat Rev Rheumatol. 2019 Feb;15(2):77-90. doi: 10.1038/s41584-018-0123-4. PMID 30498258
- [Background] Chahla J, Dean CS, Moatshe G, Pascual-Garrido C, Serra Cruz R, LaPrade RF. Concentrated Bone Marrow Aspirate for the Treatment of Chondral Injuries and Osteoarthritis of the Knee: A Systematic Review of Outcomes. Orthop J Sports Med. 2016 Jan 13;4(1):2325967115625481. doi: 10.1177/2325967115625481. eCollection 2016 Jan. PMID 26798765
- [Background] Chu CR, Rodeo S, Bhutani N, Goodrich LR, Huard J, Irrgang J, LaPrade RF, Lattermann C, Lu Y, Mandelbaum B, Mao J, McIntyre L, Mishra A, Muschler GF, Piuzzi NS, Potter H, Spindler K, Tokish JM, Tuan R, Zaslav K, Maloney W. Optimizing Clinical Use of Biologics in Orthopaedic Surgery: Consensus Recommendations From the 2018 AAOS/NIH U-13 Conference. J Am Acad Orthop Surg. 2019 Jan 15;27(2):e50-e63. doi: 10.5435/JAAOS-D-18-00305. PMID 30300216
- [Background] Filardo G, Di Matteo B, Kon E, Dhillon MS, Patel S, Marwaha N. Platelet-rich plasma for knee osteoarthritis. Am J Sports Med. 2013 Sep;41(9):NP42-3. doi: 10.1177/0363546513502635. No abstract available. PMID 23997229
- [Background] Evans CH, Kraus VB, Setton LA. Progress in intra-articular therapy. Nat Rev Rheumatol. 2014 Jan;10(1):11-22. doi: 10.1038/nrrheum.2013.159. Epub 2013 Nov 5. PMID 24189839
- [Background] Garratt AM, Brealey S, Gillespie WJ; DAMASK Trial Team. Patient-assessed health instruments for the knee: a structured review. Rheumatology (Oxford). 2004 Nov;43(11):1414-23. doi: 10.1093/rheumatology/keh362. Epub 2004 Aug 17. PMID 15316121
- [Derived] Dulic O, Abazovic D, Matijevic S, Rasovic P, Obradovic M, Bjelobrk M, Tosic M, Lalic I, Baljak B, Milinkov M. Quality of life changes in patients suffering from knee osteoarthritis treated with bone marrow aspirate concentrate, platelet-rich plasma and hyaluronic acid injections. Regen Med. 2025 Feb-Mar;20(2-3):87-96. doi: 10.1080/17460751.2025.2472589. Epub 2025 Mar 3. PMID 40028743
- [Derived] Rasovic P, Dulic O, Lalic I, Matijevic R, Janjic N, Tosic M, Aleksandric D, Abazovic D, Miskulin M, Matijevic S, Kovacevic L. The role of osteoarthritis severity, BMI and age on clinical efficacy of bone marrow aspirate concentrate in the treatment of knee osteoarthritis. Regen Med. 2023 Sep;18(9):735-747. doi: 10.2217/rme-2023-0042. Epub 2023 Aug 14. PMID 37577967
- [Derived] Dulic O, Lalic I, Kecojevic V, Gavrilovic G, Abazovic D, Miskulin M, Maric D, Bumbasirevic M. Do knee injection portals affect clinical results of bone marrow aspirate concentrate injection in the treatment of osteoarthritis? A prospective randomized controlled study. Regen Med. 2020 Aug;15(8):1987-2000. doi: 10.2217/rme-2020-0020. Epub 2020 Nov 5. PMID 33151802